CLINICAL TRIAL: NCT04917354
Title: iBEAM-Based Superb Micro-vascular Imaging for Evaluation of Hepatic Lesions
Brief Title: Superb Micro-vascular Imaging for Evaluation of Hepatic Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-025
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Hepatic Lesion
Keywords: Superb Micro-vascular Imaging; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- hepatic lesion
  Interventions: Device: Superb-Microvascular imaging

INTERVENTIONS:
Device: Superb-Microvascular imaging — Device: Superb-Microvascular imaging Superb-Microvascular imaging: new sonographic software technique on ultrasonography to detect low-vascular flow without use of contrast media for ultrasonography

SUMMARY:
Superb Micro-vascular Imaging (SMI) based on the iBeam platform is used to evaluate the blood supply of solid tumors. Compared with color Doppler technology, the sensitivity, accuracy and consistency of the ability of SMI to display blood flow are evaluated. Thus, the investigators will use Superb-Microvascular imaging (SMI, Toshiba, Japan) for diagnosing hepatic lesions, which enable to detect slow micro vascular flow inside the tumor

DETAILED DESCRIPTION:
To evaluate the diagnostic accuracy of SMI (primary outcome) when applying on the hepatic lesion.

Each US findings during exam for patients with hepatic lesion were recorded by radiologist.

Sample size calculation according to the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Visible hepatic lesion on US
2. Agree to participate in the study
3. Accessible follow-up imaging or pathological results

Exclusion Criteria:

1. Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consisted of patients (age:18-80 years) with visible hepatic lesion on US
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy | 1 week preoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- The second affilliated hospital of Zhejiang University school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No